CLINICAL TRIAL: NCT06558435
Title: Translation and Validation of "The Boston Residue and Clearance Scale" to European Portuguese
Brief Title: Validation of BRACS to European Portuguese
Status: Completed | Type: Observational
Sponsor: Centro Hospitalar de Entre o Douro e Vouga (Other)
Responsible Party: Principal Investigator, Daniela Ferreira, Speech and Language Pathologist Daniela Ferreira, Centro Hospitalar de Entre o Douro e Vouga
Other Study IDs: 252023
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Deglutition Disorders; Swallowing Disorder; Dysphagia, Oropharyngeal
Keywords: Swallowing Disorders; Dysphagia; Fiberoptic Endoscopic Evaluation of Swallowing
MeSH Terms: conditions — Deglutition Disorders | interventions — Fees and Charges

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: FEES — Single group
  Other Names: Fiberoptic Endoscopic Evaluation of Swallowing

SUMMARY:
The goal of this observational study is to translate and validate the fiberoptic endoscopic evaluation of swallowing scale "The Boston Residue and Clearance Scale - BRACS" to European Portuguese

DETAILED DESCRIPTION:
The Boston Residue and Clearance Scale (BRACS) is a multidimensional scale developed and validated to assess the severity of residues observed during fiberoptic endoscopic evaluation of swallowing (FEES).

It differs from other FEES residue scales, since it considers all aspects related to pharyngolaryngeal residues, specifically, the location, amount and the patient's clearance ability.

The purpose of this study was to translate and cross-culturally adapt the English version of the BRACS into European Portuguese and to investigate the reliability and validity of the translated version of the scale.

ELIGIBILITY:
Inclusion Criteria:

* FEES recording that allowed good visualisation of the pharynx and larynx.
* FEES recording of patients after head and neck surgery who had anatomical alterations of the structures, but which did not interfere with good visualisation of the residues.
* FEES recording of patients with a tracheostomy or under tube feeding.

Exclusion Criteria:

* FEES recording of patients under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neurological or mechanical dysphagia who have undergone a FEES examination and whose test meets the inclusion criteria described above.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Reliable and validated European Portuguese version of the BRACS | patients with neurological and/or mechanical oropharyngeal dysphagia evaluated FEES up to 3 months after the first symptomatology
  Demonstrating the reliability and validity of the Boston Residue and Clearance Scale in diagnosing dysphagia during fiberoptic endoscopic assessment of swallowing examination. BRACS it's an 11-point ordinal residue classification scale that assesses 3 aspects: the amount and location of pharyngolaryngeal residues, the presence of spontaneous swallowing to clear it and the effectiveness of patient's swallowing.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar de Entre Douro e Vouga, Santa Maria da Feira, Portugal